CLINICAL TRIAL: NCT05045651
Title: The Incidence of Anterior Knee Pain Between Unisex Knee Prosthesis and Gender Specific Knee Prosthesis Following Minimally Invasive Surgery Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Anterior Knee Pain Between Unisex Knee Prosthesis VS Gender Specific Knee Prosthesis Following MIS TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Boonchana Pongcharoen, Associated professor, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTU-EC-OT-1-005/55
Record Dates: First submitted 2021-08-29; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Osteo Arthritis Knee; Knee Pain Chronic
Keywords: anterior knee pain; gender knee prosthesis; patellar tracking; unisex knee prosthesis; total knee arthroplasty; patellar resurfacing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient specific knee prosthesis (Experimental): TKA with Gender Solution® posterior stabilized NexGen® LPS Hi-Flex; Zimmer Biomet, Inc, Warsaw, IN, USA
  Interventions: Procedure: Gender Solution®posterior stabilized NexGen® LPS Hi-Flex; Zimmer Biomet, Inc, Warsaw, IN, USA and standard posterior stabilized NexGen® LPS Hi-Flex; Zimmer Biomet, Inc, Warsaw, IN, USA
- Unisex knee prosthesis (Experimental): TKA with posterior stabilized NexGen® LPS Hi-Flex; Zimmer Biomet, Inc, Warsaw, IN, USA
  Interventions: Procedure: Gender Solution®posterior stabilized NexGen® LPS Hi-Flex; Zimmer Biomet, Inc, Warsaw, IN, USA and standard posterior stabilized NexGen® LPS Hi-Flex; Zimmer Biomet, Inc, Warsaw, IN, USA

INTERVENTIONS:
Procedure: Gender Solution®posterior stabilized NexGen® LPS Hi-Flex; Zimmer Biomet, Inc, Warsaw, IN, USA and standard posterior stabilized NexGen® LPS Hi-Flex; Zimmer Biomet, Inc, Warsaw, IN, USA — gender specific knee prosthesis:design for female to restore Q-angle, reduce anteroposterior (AP)/mediolateral(ML) ratio for reducing overhang of femoral component, increase valgus angle of trochlea groove, and reduce thickness of anterior part of prosthesis for prevention overstuff with patella. The standard TKA or unisex knee prosthesis was design for female and male.

SUMMARY:
Unisex knee prosthesis and patient specific knee prosthesis has the same anterior knee pain and patellar tracking

DETAILED DESCRIPTION:
Background:The anterior knee pain (AKP) is one of major problem of TKA. The incidence of anterior knee after TKA was 4% to 49%. The cause of AKP after TKA from surgical technique errors including joint line elevation, instability, malalignment of prosthesis, and maltracking of patella. However, AKP still has presented even high volume surgeon that prosthesis had good alignment and good stability, one of the risk factor is female. Due to female has higher Q-angle, greater anteroposterior (AP)/mediolateral(ML) ratio, smaller anterior condyle, and trochlea has higher degree of valgus angle than male. Therefore, female should has AKP even surgery with good surgical technique. The gender specific knee prosthesis was design for female to restore Q-angle, reduce anteroposterior (AP)/mediolateral(ML) ratio for reducing overhang of femoral component, increase valgus angle of trochlea groove, and reduce thickness of anterior part of prosthesis for prevention overstuff with patella. For these reasons, the gender specific knee prosthesis should reduce AKP and improve patellar tracking in female. And there is no study to compare AKP and patellar tracking between Unisex knee prosthesis and gender specific knee prosthesis following minimally invasive surgery (MIS) TKA.

Investigators asked whether AKP and patellar tracking differ between unisex knee prosthesis and gender specific knee prosthesis following MIS TKA with patellar resurfacing.

Methods:The participants were randomized into 2 groups (Gp) with computer program to make a list of random numbers of participant. Gp1 was gender specific knee prosthesis; consisted of 40 participants (40 knees) and Gp2 was unisex knee prosthesis; consisted of 40 participants (40 knees). The sample size was calculate base on anterior knee pain after TKA with a risk difference of 27% (3% versus 20%) (1,3). The 40 participants from each group would have 90% power at the 5% significant level.

Patrticipants were follow up at 2 wks, 6 wks, 3 mo, 6mo, 1 year and 2 years. At each follow up, the % anterior knee pain, VAS for anterior knee pain were record. The knee society score also was recorded and compared between two group.

All participants were operated with same surgeon and same instrumentation.

ELIGIBILITY:
Inclusion Criteria:

Aymptomatic knee OA with

* varus deformity < 30 degrees
* range of motion > 90 degrees
* flexion contracture < 20 degrees
* recurvatum < 20 degrees

Exclusion Criteria:

* gout
* postraumatic arthritis
* osteonecrosis of knee
* inflammatory joint disease

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
anterior knee pain | 4 years
  Visual analog scale for pain ( 0= no pain to 10= maximum pain), incidence for anterior knee pain (percent)
patellar tracking | 4 years
  patellar tilt > 5 degrees and/or patellar shift> 5 mm= patellar maltracking

SECONDARY OUTCOMES:
clinical outcome score | 4 years
  knee society score (0-20= poor outcomes, 21-40=fair outcomes, 41-60= good outcomes, 61-80= very good outcomes, 81-100= excellent outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Boonchana Pongcharoen, MD, Principal Investigator — faculty of medicine, Thammasat university

IPD SHARING:
Plan to Share IPD: No